CLINICAL TRIAL: NCT03967639
Title: Retrospective Analysis of Seasonal Trends of Respiratory Morbidity in Diabetic Patients
Brief Title: Seasonal Trends of Respiratory Morbidity in Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Szeged University (Other)
Collaborators: Hungarian Basic Research Council (Other); GINOP (Unknown)
Responsible Party: Principal Investigator, Barna Babik, Professor, MD, PhD, Szeged University
Other Study IDs: WHO2788-c
Record Dates: First submitted 2019-02-04; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus; Respiratory Complication; Perioperative/Postoperative Complications
Keywords: cardiac surgical procedures; respiratory mechanics; seasonal variation
MeSH Terms: conditions — Diabetes Mellitus; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group T2DM: Patients with diabetes mellitus undergoing elective cardiac surgery
  Interventions: Procedure: Elective cardiac surgery
- Group Ctrl: Control patients undergoing elective cardiac surgery without T2DM
  Interventions: Procedure: Elective cardiac surgery

INTERVENTIONS:
Procedure: Elective cardiac surgery — Elective cardiac surgery

SUMMARY:
Type 2 diabetes mellitus (T2DM) poses a significant burden on the patients and the health care system. The increasing number of surgery performed in elderly population results in an increased number of perioperative T2DM-related adverse effects. T2DM has a prevalence of 30-40% in a population undergoing cardiovascular surgery. Cardiac surgery, especially cardiopulmonary bypass (CPB) is also known to deteriorate respiratory mechanics.

Therefore, the study is aimed at a retrospective analysis of seasonal trends in respiratory consequences of T2DM, i.e.: i: distribution of patients with and without T2DM presenting for elective cardiac surgery during the two-year examination period; ii: characterization of respiratory co-morbidities in the patients, iii: exploring whether the respiratory mechanics at presentation and those caused by cardiac surgery exhibit different trends in T2DM and control patients.

DETAILED DESCRIPTION:
Our study is a retrospective analysis of patient records from all patients undergoing elective cardiac surgery between January 2007 to December 2018 at the Second Department of Internal Medicine and Cardiology Centre Cardiac Surgical Unit, University of Szeged.

Electronic and paper documentation will be examined and anonymously analysed for the following information:

1. date of cardiac surgery,
2. type of cardiac surgery procedure,
3. demographic data (age, height, weight),
4. presence of T2DM (previous diagnosis, fasting plasma glucose level, glycated haemoglobin [HbA1C]),
5. presence of respiratory co-morbidities (e.g. asthma, COPD, etc.),
6. presence of other circulatory co-mobidities (e.g. hypertension, previous stroke, vascular stenosis)

6. respiratory mechanical parameters before and after cardiac surgery, 7. presence of perioperative respiratory complications, 8. history of smoking 9. blood gas measurements before, during and after surgery

Time series statistical analysis of all data will be carried out to discover the presence of seasonal trends in both diabetic and control patients. Analysis of variance (ANOVA) will be carried out to explore global differences between diabetic and control patients.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing cardiac surgery with or without diabetes mellitus, age between 18-85 years during the time period January 2007 to December 2018

Exclusion Criteria:

* patients older than 85 years
* patients younger than 18 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of patient records from all patients undergoing elective cardiac surgery between January 2007 to December 2018 at the Second Department of Internal Medicine and Cardiology Centre Cardiac Surgical Unit, University of Szeged
Sampling Method: Probability Sample
Enrollment: 9838 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Seasonal variation in the incidence of diabetic patients undergoing cardiac surgery | Retrospective data analysis (2006-2018)
  All patient data from the time period 2006-2018 will be retrospectively analysed to explore the seasonal trends of diabetic patients (Type 1 and Type 2) undergoing cardiac surgery at a university hospital setting.
  The relative incidence of diabetic patients will be evaluated on a monthly basis in the study period.
Anthropometric data of patients undergoing cardiac surgery | Retrospective data analysis (2006-2018)
  All patient data from the time period 2006-2018 will be retrospectively analysed to explore the seasonal trends of diabetic patients (Type 1 and Type 2) undergoing cardiac surgery at a university hospital setting.
  Anthropometric data will be collected from the patient records: height (meters) and weight (kilograms) of each patient will be collected from the hospital medical records, then these data will be combined to report BMI (kg/m^2).
Comorbidities of diabetic patients undergoing cardiac surgery | Retrospective data analysis (2006-2018)
  All patient data from the time period 2006-2018 will be retrospectively analysed to explore the seasonal trends of diabetic patients (Type 1 and Type 2) undergoing cardiac surgery at a university hospital setting.
  Co-morbidities (COPD, asthma, hypertension, etc.) of each patient will be collected from the hospital medical records.
Smoking habits of patients undergoing cardiac surgery | Retrospective data analysis (2006-2018)
  All patient data from the time period 2006-2018 will be retrospectively analysed to explore the seasonal trends of diabetic patients (Type 1 and Type 2) undergoing cardiac surgery at a university hospital setting.
  Reported smoking habits (present smoker/previous smoker/never smoker; number of packs / day; duration) of each patient will be collected from the hospital medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Barna Babik, MD, PhD, Principal Investigator — Szeged University
Locations (1):
- Cardiology Centre Cardiac Surgical Unit and Second Department of Internal Medicine, University of Szeged, Szeged, Csongrád megye, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Petak F, Kovacs BN, Agocs S, Virag K, Nyari T, Molnar A, Sudy R, Lengyel C, Babik B. Seasonal changes in proportion of cardiac surgeries associated with diabetes, smoking and elderly age. PLoS One. 2022 Sep 22;17(9):e0274105. doi: 10.1371/journal.pone.0274105. eCollection 2022. PMID 36136994